CLINICAL TRIAL: NCT05221125
Title: Pilot Study of an Innovative Model to Provide Evidence-Based Multimodal Management of Neck and Back Pain in the Emergency Department (Multi-ED)
Brief Title: Multimodal Management of Neck and Back Pain in the Emergency Department (Multi-ED)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00110289
Record Dates: First submitted 2022-01-31; First posted 2022-02-02 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychologically-Informed Physical Therapy (PIPT) (Experimental): CBT-trained physical therapist evaluation and treatment with recommendation for Spine Health follow up after ED discharge
  Interventions: Behavioral: Psychologically-Informed Physical Therapy (PIPT)
- Control (No Intervention): Usual care only

INTERVENTIONS:
Behavioral: Psychologically-Informed Physical Therapy (PIPT) — The PIPT group will receive evaluation and treatment based on the PT's assessment of the individual patient's clinical presentation and condition.
  Arms: Psychologically-Informed Physical Therapy (PIPT)

SUMMARY:
The purpose of this study is to assess the feasibility and acceptability of psychologically-informed physical therapy (PIPT) in the ED in a pilot study of ED patients with neck or back pain. We will conduct a single-site, prospective trial comparing the combined program in one group with a usual care-only group. Primary outcomes will focus on feasibility based on recruitment and retention rates, and acceptability based on a 5-point patient satisfaction scale, while secondary outcomes will include pain severity, pain interference, anxiety, physical function, opioid use, repeat ED visits, and hospitalizations at 1 hour and at 24 hours, 1 month and 3 months after ED discharge.

We will use pilot study results to develop a protocol for a larger pragmatic randomized clinical trial designed to rigorously evaluate PIPT in the ED combined with Spine Health follow up for ED patients with neck or back pain. We will perform a process evaluation of our proposed clinical trial study design, including characterizing and quantifying the degree of CBT and PT components used by treating PTs while in the ED and during Spine Health follow up, number of Spine Health visits attended in the first month, and integration into usual ED care. Qualitative interviews will be used to identify facilitators, barriers and potential solutions to intervention and research study procedures based on the patients' experience.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 18 years or older),
* Presented to the ED with pain in the neck and/or back,
* A diagnosis of musculoskeletal pain as determined by an ED provider,
* Able to read and understand the consent form in English.

Exclusion Criteria:

* Suspected to have a non-musculoskeletal cause of pain;
* Unable to provide informed consent or to comprehend or complete study measures or procedures due to cognitive impairment, including evidence of drug, medication or alcohol intoxication, or due to severe hearing or speech impairment;
* Unable to safely participate due to critical illness, emergent surgical need, other serious medical condition (including active COVID-19 infection),
* ED provider judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Number of ED patients eligible for recruitment as measured by patient log | Post implementation, up to 6 weeks
Number of patients enrolled as measured by patient log | Post implementation, up to 6 weeks
Number of patients retained in study as measured by patient log | Post implementation, up to 6 weeks
Number of patients that found treatment satisfactory via satisfactory questionnaire | Post implementation, up to 6 weeks
  5 point Likert-scale satisfaction scale

SECONDARY OUTCOMES:
Change in Pain Score | ED pre-treatment (baseline); ED post-treatment (1 hour); 24 hours post discharge
  11-point Numeric Rating Scale (NRS) for current pain
Change in Anxiety Level | ED pre-treatment (baseline); ED post-treatment (1 hour); 24 hours post discharge
  Subjective Units of Discomfort Scales (SUDS)
Change in Function | ED pre-treatment (baseline); ED post-treatment (1 hour); 24 hours post discharge
  PROMIS-29
Change in Quality of Life (QoL) | ED pre-treatment (baseline); ED post-treatment (1 hour); 24 hours post discharge
  PROMIS-29
Change in pain related distress | ED pre-treatment (baseline); 1 and 3 months post discharge
  Optimal Screening for Prediction of Referral and Outcome (OSPRO) tool
Change in self efficacy | ED pre-treatment (baseline); 1 and 3 months post discharge
  Optimal Screening for Prediction of Referral and Outcome (OSPRO) tool
Change in severity of chronic pain | ED pre-treatment (baseline); 1 and 3 months post discharge
  Simplified graded chronic pain scale
Number of pain medications prescribed | up to 3 months post discharge
  as measured by chart review
Number of Spine Health referrals for follow up PT | At ED discharge (up to 48 hours)
  as measured by chart review
Number of Spine Health visits for follow up PT | up to 3 months post discharge
  as measured by chart review
Number of repeat ED visits | up to 3 months post discharge
  as measured by chart review
Number of patient hospitalizations | up to 3 months post discharge
  as measured by chart review

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Eucker, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Hospital Emergency Department, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No